CLINICAL TRIAL: NCT02837276
Title: Intermittent Hypoxemia and Acute Kidney Injury Study (IHAKI Study)
Acronym: IHAKI
Status: Completed | Type: Observational
Sponsor: Elie G. Abu Jawdeh, MD (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Elie G. Abu Jawdeh, MD, Assistant Professor of Pediatrics, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 13-0232-F1V
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Intermittent Hypoxemia; Acute Kidney Injury; Preterm Infant
Keywords: Intermittent Hypoxemia; Acute Kidney Injury; Preterm infant
MeSH Terms: conditions — Acute Kidney Injury; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pilot study aims at investigating the relationship between intermittent hypoxemia (IH) and acute kidney injury (AKI) in preterm infants.

AIM 1: Test the hypothesis that intermittent hypoxemia is associated kidney injury in preterm infants, as reflected by a rise in serum creatinine.

AIM 2: Test the hypothesis that there is rise in acute kidney injury urinary biomarkers with increased intermittent hypoxemia.

DETAILED DESCRIPTION:
BACKGROUND:

Preterm birth is a major health care concern and although survival of premature infants has improved, the incidence of neonatal morbidities has slightly decreased especially in cases of extreme prematurity. Apnea of prematurity (immature respiratory control) is a major complication in Neonatal Intensive Care Units occurring in virtually all infants born before 28 weeks gestation. Intermittent Hypoxemia (IH), episodic oxygen desaturation events, is generally attributed to apnea of prematurity often superimposed upon suboptimal lung function. Intermittent hypoxemia events are common in preterm infants and may lead to both short-term and long-term morbidities. Typically, the incidence of intermittent hypoxemia (IH) increases over the first 4 weeks of life before plateauing at weeks 6-8. In addition to inducing oxidative stress by increasing production of reactive oxygen species, this hypoxemia/reoxygenation cycle is thought to induce a pro-inflammatory cascade of transcription factors that promotes activation of inflammatory cells resulting in multisystem morbidity. These morbidities include retinopathy of prematurity, cardiorespiratory instability, and poor neurodevelopmental outcomes. A potential morbidity that has yet to be investigated is acute kidney injury (AKI).

AKI is associated with morbidity and mortality in critically ill neonates. The risk of AKI is higher in very low birth weight infants requiring assisted ventilation and ionotropic support, and in infants with congenital heart disease. Additionally, AKI occurs more frequently in infants who suffered severe birth asphyxia. While it has been established that end-stage kidney disease (ESKD) is associated with worsening sleep apnea in adults, it has been proposed that sleep apnea and nocturnal hypoxemia may contribute to kidney injury, the development of chronic kidney disease (CKD), and the progression to kidney failure. Proposed mechanisms of kidney disease via intermittent nocturnal hypoxemia include 1: direct intrarenal hypoxemia (resulting in tubulointerstitial injury) 2: an increase in oxidative stress, inflammatory cytokines, and systemic blood pressure (via activation of the renin-angiotensin system). Hence It is plausible that IH may modulate AKI in preterm neonates. The investigators goal is to test the hypothesis that intermittent hypoxemia is associated with Acute Kidney Injury in preterm infants. Investigation of relationship between IH and AKI may provide further insight into onset and prevention given the recent advancements in the detection and characterization of AKI in this vulnerable population.

SPECIFIC AIMS:

AIM 1: Test the hypothesis that intermittent hypoxemia is associated kidney injury in preterm infants, as reflected by a rise in serum creatinine.

APPROACH: Premature infants with GA 23 to 31 weeks will be prospectively recruited from Kentucky Children's Hospital Neonatal Intensive Care Unit (NICU). High resolution oxygen saturation monitoring will be performed for the first 2 months of life. Creatinine levels will be collected as they are obtained routinely on premature infants in the NICU. Demographic data will be collected including gestational age, postnatal age, gender and race. Clinical data including respiratory support, caffeine use, vital signs and neonatal morbidities will be documented. Scores to predict severity of disease and mortality in newborns will be used. The investigators will assess the cumulative effect of IH on AKI as reflected by serum creatinine measurements at 1 month, 2 months, and discharge in extremely preterm infants.

AIM 2: Test the hypothesis that there is rise in acute kidney injury urinary biomarkers with increased intermittent hypoxemia.

APPROACH: Similar to Aim 1, premature infants with GA 23 to 31 weeks will be prospectively recruited from Kentucky Children's Hospital Neonatal Intensive Care Unit (NICU). High resolution oxygen saturation monitoring will be performed for the first 2 months of life. Urine will be collected daily in the first week of life and then weekly until 2 months of age and hospital discharge. Collecting urine is noninvasive and minimal risk. Samples will be de-identified and stored in the investigators research laboratory. Standardized kits to measure biomarkers associated with kidney injury such as albumin, β2-microglobulin (β2MG), cystatin C (Cys C), epidermal growth factor (EGF), neutrophil gelatinase associated lipocalin (NGAL), osteopontin (OPN), and uromodulin (UMOD) will be used. Since IH increases with age and persists during NICU stay, the cumulative effect of intermittent hypoxemia will be correlated with biomarker concentrations weekly throughout the study period and at discharge.

Oxygen saturation will be continuously monitored upon admission with high resolution pulse oximeters, with 2 second averaging time and 1Hz sampling rate. Novel software will be utilized to analyze raw data per the following definitions:

1. Intermittent Hypoxemia is primarily defined as a drop in oxygen saturation (SpO2) to less than 80% for more than 4 seconds and less than 3 minutes.

   Secondary measures for IH include:
2. A drop in SpO2 of <85% for >4 seconds and <3 minutes duration
3. A decline in SpO2 by >4% from baseline to <90% that lasted >4 seconds
4. Percent time spent below above threshold, includes sustained hypoxemia (>3min duration)
5. Number of hyperoxemic events defined as an increase in SpO2 of >95%
6. Duration and nadir of each oxygen desaturation and hyperoxemic event
7. Mean SpO2/day

Sample size: There is no data available in the literature to calculate sample size. Based on NICU census, consent success rate, and accounting for data loss, the investigators will recruit a total of 50 patients for this pilot project. To maintain a balanced sample, the investigators will stratify enrollment by gestational age targeting 15-18 subjects in each of the following groups: 23-25 weeks gestation, 26-28 weeks gestation, 29-31 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than 32 weeks gestational age admitted to University of Kentucky neonatal intensive care unit

Exclusion Criteria:

* Major congenital malformations

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants less than 32 weeks gestational age.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that intermittent hypoxemia is associated with acute kidney injury, as reflected by a rise in creatinine or urinary biomarkers | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elie G Abu Jawdeh, MD, Principal Investigator — University of Kentucky; Mina H Hanna, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky - Kentucky Children's Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No